CLINICAL TRIAL: NCT03293368
Title: Efficacy of Intralesional Injection of Autologous Platelet Rich Plasma Versus Intralesional Injection of Corticosteroids on Pain Relief and Ulcers Healing in Patients With Erosive Oral Lichen Planus; Randomized Clinical Trial
Brief Title: Efficacy of Intralesional Injection of Platelet Rich Plasma in the Treatment of Patients With Erosive Oral Lichen Planus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelhameed Hamid Mohammad Hijazi, PhD Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP-olp
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Erosive Oral Lichen Planus
Keywords: Oral; Lichen planus; PRP
MeSH Terms: conditions — Lichen Planus | interventions — Intercellular Signaling Peptides and Proteins; Triamcinolone Acetonide; Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (Experimental): 0.5 ml of autologous platelet rich plasma prepared using a double spin technique described by Mostafa et al., 2013 will be injected in the center of eroded oral mucosa in patients suffering from oral lichen planus.
  Interventions: Biological: Platelet rich plasma
- Croticosteroids (Active Comparator): 0.5 ml of triamcinolone acetonide 40 mg will be injected in the center of eroded oral mucosa in patients suffering from oral lichen planus.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Biological: Platelet rich plasma — Platelet rich plasma will be prepared from the patients own blood in the same visit using a double spin technique, then 0.5 ml of PRP will be injected per 1 cm2 of eroded oral mucosa.
  Other Names: Platelet rich in growth factors
  Arms: Platelet rich plasma
Drug: Triamcinolone Acetonide — 0.5 ml of triamcinolone acetonide 40mg will be injected per 1 cm2 of eroded oral mucosa
  Other Names: Corticosteroids, Steroids
  Arms: Croticosteroids

SUMMARY:
After signing the informed consent, the participant will be allocated to either intervention or control group, then each participant in the intervention group will receive intralesional injections of platelet rich plasma extracted from their own blood in each visit as following:

1. 12 ml of blood will be assembled from the veins of antecubital fossa
2. PRP preparation will be done according to Mostafa et al., 2013
3. 0.5 ml of PRP will be injected per 1 cm2 of ulcerated mucosa

The second group will receive triamcinolone acetonide 40 mg injected 1 ml per 1 cm2 of ulcerated mucosa

Both groups will receive a total of 4 injection, the injections will be carried out once a week.

Pain, lesions size and remission time are the outcomes will be assessed using a numerical rating scale (Seymour, 1982), clinical score according to Thongprasom et al., 1992 and binary scale for remission time according to Conrotto et al., 2006, respectively.

Assessment of the outcomes will be carried before the trial (baseline records) and before receiving the treatment in each visit by the primary investigator (H.A.) and the blinded assessor (Dr. A.W.) separately.

Each participant will have a total of 11 visits during the trial, 5 visits will be once every week during the trial and every 2 weeks for 3 months treatment free.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with a clinical picture that assumes the diagnosis of erosive oral lichen planus (bilateral, more or less symmetrical erosive lesions with lacelike network of slightly raised gray white lesions (reticular pattern), and a histological findings that confirms the diagnosis (liquefaction degeneration of the basal cell layer with irregular-saw teeth like rete pegs.

Exclusion Criteria:

* Systemic disorders such as hematological diseases, severe cardiovascular diseases, treatment with any drugs that could cause Lichenoid reaction.
* Pregnancy or active breastfeeding
* Patients who had lesion/lesions with dysplasia
* Patients who received topical treatment for Oral Lichen planus in the last 2 weeks (Lee et al., 2013) or systemic treatment for OLP in the past 3 months.
* Platelet count < 150,000/mm3; Hgb < 11 g/dl.
* Immunosuppressed patients
* Patients receiving therapy with anticoagulants and use of non-steroidal anti-inflammatory drugs in the 5 days before taking the blood sample.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Reported Pain | 3 months
  Pain and burning sensation assessed using Numerical rating scale

SECONDARY OUTCOMES:
Clinical score | 3 months
  Clinical score using a 5 grades scoring system described by Thongprasom et al.,1992
Remission time | 3 months
  Time until flare up of the disease occur using a binary scale (Stable/Not stable) described by Conrotto et al., 2006

CONTACTS AND LOCATIONS:
Overall Officials: Soheir Gaafar, Professor, Study Chair — Professor of oral medicine, diagnosis and periodontology. Faculty of Dentistry. Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hijazi A, Ahmed W, Gaafar S. Efficacy of intralesional injections of platelet-rich plasma in patients with oral lichen planus: A pilot randomized clinical trial. Clin Exp Dent Res. 2022 Jun;8(3):707-714. doi: 10.1002/cre2.550. Epub 2022 Feb 26. PMID 35218680

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/68/NCT03293368/Prot_SAP_000.pdf